CLINICAL TRIAL: NCT06456424
Title: Bacteriophage Therapy for Methicillin-Sensitive Staphylococcus Aureus Prosthetic Joint Infection
Acronym: PHAGE-2024-01
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: University of Toronto (Other); Precisio Biotix Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB23-1733; Control #: 286405 (Other: Health Canada); Dossier ID: HC6-024-c283712 (Other: Health Canada)
Record Dates: First submitted 2024-05-29; First posted 2024-06-13 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Prosthetic Joint Infections of Hip; Staphylococcus Aureus Infection
Keywords: Single patient; Bacteriophage; Phage
MeSH Terms: conditions — Staphylococcal Infections | interventions — Phage Therapy

STUDY DESIGN:
Intervention Model Description: Single patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open Label Arm (Experimental): Bacteriophage cocktail
  Interventions: Biological: Phage therapy

INTERVENTIONS:
Biological: Phage therapy — Bacteriophage cocktail consisting of phages BP13 and J1P3

SUMMARY:
This is a single-patient, phase I/II clinical trial that aims to evaluate the potential of a bacteriophage cocktail to treat and prevent the recurrence of a methicillin-susceptible Staphylococcus aureus prosthetic joint infection of the hip. The patient has exhausted all conventional therapies, both surgical and medical, at considerable detriment to his quality of life. The treatment involves a one time, intra-operative injection of bacteriophages into the joint and 14 days of intravenous phage therapy. The goal is to eliminate the infection and prevent further complications, providing a potential new treatment avenue for patients with difficult-to-treat infections.

DETAILED DESCRIPTION:
This study is a single-patient, phase I/II clinical trial that addresses a challenging case of a recurrent methicillin-sensitive Staphylococcus aureus (MSSA) infection in a prosthetic hip joint despite extensive antibiotic treatments and multiple surgeries.

Given the failure of conventional treatments and the high risk associated with major surgical interventions, this study explores the use of bacteriophage therapy as an innovative alternative. Bacteriophages, viruses that specifically infect and lyse bacterial cells, offer a patient-specific, targeted approach to combating bacterial infections within biofilms. Our study will use a bacteriophage cocktail containing phages BP13 and J1P3, both of which have demonstrated in-vitro activity against the patient's strain of S. aureus.

The treatment protocol involves the administration of phages intra-articularly on day 1 and intravenously twice daily on days 1-14. This dual approach aims to enhance the efficacy of the phage therapy by ensuring both systemic and localized delivery of the phages to the infected site.

The primary outcome will be the resolution of the infection, indicated by the absence of clinical symptoms such as wound drainage, swelling, erythema, pain, and fever, as well as the normalization of inflammatory markers over a 12-month period following the phage therapy.

Throughout the study, the patient's safety and response to the treatment will be rigorously monitored through regular physical examinations, blood tests, and if needed, imaging studies. The initial dose of the phage cocktail will be administered in a hospital setting to monitor for any immediate adverse reactions Follow-up assessments will continue for a year to ensure long-term efficacy and safety.

The goal of this study is to demonstrate the potential of bacteriophage therapy as a viable treatment option for prosthetic joint infections, particularly those resistant to standard treatments. Success in this case could pave the way for broader applications of phage therapy in managing complex bacterial infections, offering a new avenue for treatment where traditional methods have failed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of active chronic prosthetic joint infection
* Causative bacteria is susceptible to bacteriophage therapy in vitro
* History of multiple failed antibiotic and surgical interventions

Exclusion Criteria:

* Stage 5 chronic kidney disease
* Cirrhosis
* A known allergy to phage products
* Fever
* Involvement in another clinical trial
* Pregnancy

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Clinical response | 1 year
  Resolution of the infection, indicated by the absence of clinical symptoms such as wound drainage, swelling, erythema, pain, and fever. This will be determined by a questionnaire and monthly assessments by a Infectious Disease physician.

SECONDARY OUTCOMES:
Safety of phage therapy | 29 days
  The safety outcome focuses on monitoring and documenting any adverse events (both serious and not) or reactions associated with bacteriophage therapy. Key safety measures include observing for immediate allergic reactions during the first dose, conducting regular clinical assessments, and performing routine blood tests (complete blood counts, lymphocyte subsets, c-reactive protein, liver function tests, serum electrolytes and serum creatinine) to detect any potential organ damage or unexpected side effects.
Microbiologic response | 1 year
  Bacterial cultures from the infected joint will be sent on an as-needed basis should the patient develop another draining fistula or require a repeat surgical incision and drainage. If there is no need to send bacterial cultures, or if bacteria other than Staphylococcus aureus are isolated, then this would be a good microbiologic response.
Biochemical response | 1 year
  To monitor for subclinical infection the patient will have serum inflammatory markers (white blood cell count and c-reactive protein) sent on days 0, 2, 4, 8, 11, 15, 29, and then every 30 days afterwards. Should both inflammatory markers decrease to be within the normal limits this would be a good biochemical response.

CONTACTS AND LOCATIONS:
Locations (1):
- South Health Campus, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No